CLINICAL TRIAL: NCT06860373
Title: LIFE-DSR-Biomarker Sub-study of Biomarkers in Down Syndrome Related Alzheimer's Disease (DS-AD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to recruit
Sponsor: LuMind IDSC Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LIFE-DSR-BIO DS-AD
Record Dates: First submitted 2024-03-22; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-06

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Masking Description: There is no masking for this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiotracer [18F]MK-6240 (Other): In this sub-study, participants will have two [18F]MK-6240 tau PET scans. Participants will undergo administration of [18F]MK-6240 to detect the presence of tau in the brain. The applied [18F]MK-6240 radioactive dose will be approximately 5 mCi (185 MBq) ± 20%. The mass dose will not exceed 20 µg. This is the only arm.
  Interventions: Biological: [18F]MK-6240

INTERVENTIONS:
Biological: [18F]MK-6240 — [18F]MK-6240 will be synthesized, purified, and formulated at the local radiochemistry synthesis laboratory and will be administered as a sterile, pyrogen-free solution by IV injection.

SUMMARY:
This is an optional sub-study that will enroll participants from the LIFE-DSR parent protocol. Participants will undergo assessments at two timepoints, including: additional blood samples for PBMC and RNA extraction, as well as a lumbar puncture for collection of CSF, and/or MRI and tau PET imaging. Sub-study visits will be scheduled around a similar calendar-day as the parent protocol study visits (e.g., Month (M) 0 (M0) and M16, or M16 and M32).

DETAILED DESCRIPTION:
This is an optional sub-study that will enroll participants from the LIFE-DSR parent protocol. Participants will undergo assessments at two timepoints, including: additional blood samples for PBMC and RNA extraction, as well as a lumbar puncture for collection of CSF, and/or MRI and tau PET imaging. Sub-study visits will be scheduled around a similar calendar-day as the parent protocol study visits (e.g., Month (M) 0 (M0) and M16, or M16 and M32).

The aim is to increase knowledge of biomarkers of interest in DS-AD clinical progression and perform deep immunophenotyping of PBMC samples. Intervention studies in people with DS depend upon determining the optimal age for treatments to be given, by identifying or developing reliable outcome measures that are most sensitive to decline and discovering biomarkers most closely related to disease progression.

For tau deposition, the aim of this study is to ascertain the degree and distribution of tau pathology in DS as a function of age using tau PET, and to determine the longitudinal progression of that pathology. As such, enrichment of the study population included in the tau PET sub-study for presence of tau PET positive scans, and in particular tau PET scans in the earliest stages of positivity, is desirable. Accomplishing this may require flexibility in recruitment, including adjustments of age eligibility as a response to emerging new information in the sub-study population as the study proceeds. PET images will be reviewed in near real-time to enable adaption of the age strata based on the presence or absence of tau PET signal.

All the above endpoints will be acquired with informed consent and assent. All data is intended for research purposes only and associated clinical data will be stored securely.

Participants will have the option to participate in:

* LP to collect CSF and venipuncture to collect a blood sample OR
* Imaging (MRI and tau PET) and venipuncture to collect a blood sample OR
* Both

  * LP to collect CSF and venipuncture to collect a blood sample AND
  * Imaging (MRI and tau PET).

ELIGIBILITY:
Inclusion Criteria:

1. The participant must be currently enrolled in the LIFE-DSR parent protocol.
2. The adult with DS must be age 35 to 55 years.
3. Both the participant, or LAR, and their caregiver must be able to understand and be willing to provide consent. The LAR will sign the informed consent. The participant will sign the informed consent or assent.
4. Both the participant, or LAR, and their caregiver must be willing to comply with the scheduled visits and scheduled assessments.
5. Agreement of caregiver and clinician the participant can cooperate with protocol tasks.

Exclusion Criteria:

Participants meeting any of these criteria are excluded from the LP portion of the sub-study.

1. Assessment (per medical history, physical exam, vital signs or other clinically relevant measure or circumstance) which, in the opinion of the site PI, makes the participant unsuitable for participation in this study.
2. Evidence for raised intracranial pressure. Examples include papilledema on physical exam or CNS lesion with mass effect.
3. Presence of lower spinal malformations, prior lumbosacral spinal surgery, local infection, or other abnormalities that would exclude lumbar puncture.
4. Allergy to Lidocaine (xylocaine) or its derivatives.
5. Evidence or history of significant active bleeding or coagulation disorder, or use of anticoagulant medications such as coumadin, heparin, thrombin inhibitors (e.g., dabigatran) or factor Xa inhibitors (e.g., apixaban).
6. Previous or ongoing treatment with aducanumab (AduhelmTM) OR any anti-amyloid OR any anti-tau antibody OR investigational treatment within the previous 30-calendar days of this sub-study baseline LP. Treatment with AduhelmTM is permitted in the LIFE-DSR parent protocol but precludes participation in this LP sub-study.

   Participants meeting any of these criteria are excluded from the imaging portion of the sub-study.
7. Contraindication to MRI or PET scans, evidenced by presence or history of any significant or uncontrolled medical condition which, in the opinion of the Investigator, would increase the potential risk to the study participant (e.g., history of CNS infection, history of exposure to CNS toxin, epilepsy, sensitivity to flashing lights, pacemaker).
8. Participants in whom MRI is contraindicated including, but not limited to, those with a pacemaker, presence of metallic fragments near the eyes or spinal cord or cochlear implant. Dental fillings do not present a risk for MRI.
9. Suffers from claustrophobia, inability to tolerate confined spaces, or prior failed experience completing MRI scans or blood draws.
10. Positive pregnancy test or currently breast-feeding.
11. Previous or ongoing treatment with aducanumab (AduhelmTM) OR any anti-amyloid OR any anti-tau antibody OR investigational treatment within the previous 30-calendar days of this sub-study baseline PET. Treatment with AduhelmTM is permitted in the LIFE-DSR parent protocol but precludes participation in this imaging sub-study.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure to establish a biobank specifically for DS participants | Month 0 and Month 16 or Month 16 and Month 32
  CSF AD biomarkers measured longitudinally at approximately Month 0 and Month 16 or Month 16 and Month 32.
  Establish a biobank specific to DS to receive, store and distribute biospecimens supporting future Omics, biomarker analyses, epigenetic studies, and genotyping. Biomarker candidates will be determined when the study ends and may include primary analytes such as AB42, AB40, AB42/40 ratio, t-tau, p-tau, NfL.
  Evaluate prespecified CSF biomarkers using technically validated immunoassays on the Quanterix, Mesoscale and Abcam Fireplex Cytokine assay platforms. Biomarker candidates will be determined when the study ends and may include primary analytes such as AB42, AB40, AB42/40 ratio, sAPP, sAPPB, t-tau, p-tau, soluble-TREM2, NfL, GFAP, UCHL1, Tau.
Primary Outcome to ascertain the degree and distribution of tau pathology in DS as a function of age using tau PET | Month 0 and Month 16 or Month 16 and Month 32
  Burden of total and regional tau deposition, relative to baseline, as measured by [18F]MK-6240 uptake. This outcome will provide information regarding:
  Expected rates of change given baseline amyloid and tau burden, The sample sizes required to detect a reduction in the rate of accumulation at different stages of AD, and Homogeneity and heterogeneity in tau spatial distribution at different stages of AD progression.
  Correlate the tau PET imaging data with the cognitive, behavioral, functional assessments and medical history data collected in the LIFE-DSR parent protocol to better establish the stage of AD for each participant.

SECONDARY OUTCOMES:
Secondary Outcome is to increase knowledge of biomarkers of interest in DS-AD clinical progression and perform deep immunophenotyping of PBMC and plasma samples. | Month 0 and Month 16 or Month 16 and Month 32
  The secondary outcome measures include changes relative to baseline compared to AD plasma biomarkers such as A42, A40, NfL, and p-tau 217 and genetic biomarkers of risk such as APOE
  Conduct deep immunophenotyping of peripheral blood mononuclear cells (PBMCs)
  Determine within-participant and between-participant variability of specific biomarker candidates in the plasma, PBMCs, CSF and CSF resident immune cells collected at two time points approximately 16 months apart.
  Month 0 and Month 16 or Month 16 and Month 32

OTHER OUTCOMES:
Exploratory Outcome - Biomarkers Comparisons | through study completion, an average of 2 years
  The exploratory outcomes include comparisons of CSF AD biomarkers to biomarkers of other modalities (i.e., plasma biomarkers, tau PET imaging, CSF, and plasma cytokines, PBMC and CSF resident cell immunophenotypes) to determine within-participant and between-participant variability of specific biomarker candidates. The identification of specific biomarkers to be used will be determined after the study has ended.

CONTACTS AND LOCATIONS:
Locations (1):
- Barrow Neurological Institute, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided